CLINICAL TRIAL: NCT04216069
Title: Evaluation of the Efficacy of a Commercially Available Regimen Versus Brushing Alone on Established Plaque and Gingivitis on Adolescents: Study Protocol for a Randomized, Controlled, Blind Clinical Trial
Brief Title: Efficacy of Different Toothbrushes and Hygiene Regimen
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Toothbrushes
Record Dates: First submitted 2019-12-18; First posted 2020-01-02 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Dental Plaque; Halitosis
MeSH Terms: conditions — Dental Plaque; Halitosis | interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will not know to which group the participant belongs.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total 12 regimen group (Experimental): This group will use the following procedure: Colgate Ultrasoft toothbrush, Colgate Total 12 toothpaste and Plax Mouthwash.
  Interventions: Other: Total 12 regimen
- Tooth brushing alone group (Experimental): This group will use Colgate Ultrasoft toothbrush and Colgate Cavity Protection toothpaste.
  Interventions: Other: Toothbrushing alone

INTERVENTIONS:
Other: Total 12 regimen — The volunteers will be invited with their caregivers to a lecture administered with the aim of clarifying the importance of oral hygiene and motivating brushing among the volunteers. Written clarifications will also be given in the form of an illustrative pamphlet. The volunteers will be trained in the technique through supervised brushing in front of a mirror. Subjects from the Group 1 will use a regimen with Colgate Total 12 toothpaste + Plax mouthwash + Colgate Ultrasoft toothbrush. Subjects will be instructed to use only their assigned group during the study period. The treatment products will be re-supplied at regular intervals. Subjects will return with their assigned products to the study site before receiving new products.
  There will be no restrictions regarding diet habits during the course of the study. Upon completion of the study, subjects will be instructed to return all used and used products.
  Arms: Total 12 regimen group
Other: Toothbrushing alone — The volunteers will be invited with their caregivers to a lecture administered with the aim of clarifying the importance of oral hygiene and motivating brushing among the volunteers. Written clarifications will also be given in the form of an illustrative pamphlet. The volunteers will be trained in the technique through supervised brushing in front of a mirror. Group 2 will use Colgate Cavity Protection Toothpaste + Colgate Ultrasoft toothbrush. Subjects will be instructed to use only their assigned group during the study period. The treatment products will be re-supplied at regular intervals. Subjects will return with their assigned products to the study site before receiving new products.
  There will be no restrictions regarding diet habits during the course of the study. Upon completion of the study, subjects will be instructed to return all used and used products.
  Arms: Tooth brushing alone group

SUMMARY:
To evaluate: 1) Evaluate the efficacy of a regimen commercially available versus brush alone on established plaque and gingivitis on adolescents. The Group 1 will use the following procedure: Colgate Ultrasoft toothbrush, Colgate Total 12 toothpaste and Plax Mouthwash, and the other Group will use Colgate Ultrasoft toothbrush and Colgate Cavity Protection toothpaste; 2) The level of halitosis. Two calibrated and blinded examiners (Cohen Kappa 85%) will evaluate the gingival condition using the visible plaque indices, a simplified oral hygiene index - IHOS and gingival bleeding index, with the aid of a WHO probe. For the evaluation of halitosis levels, all individuals will respond to a questionnaire regarding personal data, general and oral health, which includes hygiene habits and received previous guidelines for the procedures to be performed in the second moment. At the next consultation, subjects will be assessed clinically for halitosis using the portable BreathAlert™ sulfide monitor (Tanita Corporation, Japan), in addition to the evaluation of the tongue flap index (ISL), pH and salivary flow. The evaluations will be in the following periods: baseline, 1, 3 and 6 months of brushing. Data will be submitted to descriptive statistical analysis to demonstrate the distributions frequency of biofilm indices and gingival bleeding. The differences in the criteria evaluated will be submitted to Fisher's exact test (α = 0.05) and their performance at different times will be evaluated by the Mann-Whitney test (α = 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Good general health;
* Age 12 to 17;
* Absence of motor, comprehension and cognitive difficulties that impede adequate oral hygiene.

Exclusion Criteria:

* Active dental caries with cavity exposing dentin (visible cavity) on teeth for which the simplified oral hygiene index will be used. If these teeth are not present, adjacent teeth may be considered;
* Teeth with formation defects and dental crowding;
* Periodontal disease (tooth mobility > 2 mm, pocket > 5 mm, gingivitis);
* Parafunctional habits (bruxism, nail biting), active clamps for removable partial dentures, use of orthodontic appliance;
* Volunteer or legal guardian who does not agree with the terms of the study or has difficulty appearing for the follow up appointments;
* Pregnant volunteers;
* Use of medications that alter gingival health, such as antibiotics, in the previous three months;
* Use of mouthwash or toothpaste containing products for the control of biofilm;
* Smokers;
* Systemic disease (diabetes).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2021-01-05 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-25 (Estimated)

PRIMARY OUTCOMES:
Evaluation of change in biofilm index | Baseline, after 1, 3 and 6 months of toothbrushing.
  The gingival health assessments will be performed through a visual examination for the determination of the visible plaque index, gingival bleeding and oral health at baseline as well as after the use of brush.

SECONDARY OUTCOMES:
Change in halitosis index | Baseline, after 1, 3 and 6 months of toothbrushing.
  Halitosis index using the portable BreathAlert™ sulfide monitor (Tanita Corporation, Japan).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Metropolitana de Santos, Santos, São Paulo, Brazil